CLINICAL TRIAL: NCT03398707
Title: The Impact of a Bundle of Preventive Measures for Post-intensive Care Syndrome on the Outcome of Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, Director of ICU, Hospital Sao Domingos
Other Study IDs: PICS study
Record Dates: First submitted 2017-12-24; First posted 2018-01-12 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2018-12

CONDITIONS: PICS
Keywords: PICs; diagnosis; prevention; outcome
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational cohort study will investigate the impact of a bundle of nine preventive measures (Assessment, prevention and management of pain; spontaneous awaking trial; spontaneous breathing trial; choice of sedation and analgesia; delirium assessment, prevention and management; early mobility; family communication and ICU Diary) on the incidence and severity of Post-Intensive Care Syndrome (PICS) and clinical outcomes in critically ill patients

DETAILED DESCRIPTION:
This is a prospective observational cohort study. It will include all adult patients, admitted to a surgical ICU (13 beds) and a medical ICU (10 beds), with a length of ICU stay of at least 2 day, from January 01 to December 31 2018. Patients with severe cognitive deficits prior to admission, identified by clinical history obtained by the psychology or through the Mental State Mini Exam (MMSE), traumatic brain injury and stroke patients with Glasgow coma scale <14, will be excluded. On admission to the ICU, risk factors for PICS will be identified.

During ICU stay, the patients will be submitted to nine interventions aiming at the prevention of PICS: Assessment, prevention and management of pain; spontaneous awaking trial; spontaneous breathing trial; choice of sedation and analgesia; delirium assessment, prevention and management; early mobility; family communication and ICU Diary. At ICU discharge, the physical, psychiatric and cognitive components of PICS will be evaluated using the following tools: FSS-ICU, dynamometry and nutritional indicators (physical component), HADS (Anxiety and Depression), MOCA (cognitive dysfunction) and PCL -C (posttraumatic stress disorder). The duration of mechanical ventilation, duration of sedation, ICU LOS and hospital mortality will also be evaluated. Reassessments will be done 5 days after discharge from the ICU or at hospital discharge (what happens first) and 3 months after the randomization at the follow-up clinic. Patients identified with PICS at discharge from the ICU will be compared with those who did not develop the syndrome. The investigators will specifically evaluate the percentage of adherence to preventive measures, the presence of risk factors and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria: .

* Adult non pregnant patients
* Length of ICU stay of at least 2 days.

Exclusion Criteria:

* Severe cognitive deficits prior to admission.
* Traumatic brain injury with Glasgow coma scale < 14
* Stroke with Glasgow coma scale < 14

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients, admitted to a surgical ICU (13 beds) and a medical ICU (10 beds), with a length of ICU stay of at least 2 day, from January 01 to December 31 2018. Patients with severe cognitive deficits prior to admission, identified by clinical history obtained by the psychology or through the Mental State Mini Exam (MMSE), traumatic brain injury and stroke patients with Glasgow coma scale <14, will be excluded.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive function | Change from baseline at the time of discharge from the ICU, 5 days after discharge from the ICU or at the time of hospital discharge (whichever occurs first) and after 3 months of randomization at the follow-up clinic
  Evaluation of cognitive dysfunction using the Montreal Cognitive Assessment (MOCA) tool,
Change in Psychiatric function | Change from baseline at the time of discharge from the ICU, 5 days after discharge from the ICU or at the time of hospital discharge (whichever occurs first) and after 3 months of randomization at the follow-up clinic
  Evaluation of psychiatric dysfunction using the HADS (Hospital Anxiety and Depression Scale).
Change in Post-traumatic stress syndrome | Change from baseline at the time of discharge from the ICU, 5 days after discharge from the ICU or at the time of hospital discharge (whichever occurs first) and after 3 months of randomization at the follow-up clinic
  Identification of post-traumatic stress syndrome through PCL-C (Post-traumatic stress checklist-civilian)
Change in physical function | Change from baseline at the time of discharge from the ICU, 5 days after discharge from the ICU or at the time of hospital discharge (whichever occurs first) and after 3 months of randomization at the follow-up clinic
  Evaluation of physical dysfunction through FSS-ICU (Functional status score in the ICU)

SECONDARY OUTCOMES:
The duration of mechanical ventilation, | During ICU stay.. Expected average 21 days
  The duration of mechanical ventilation in days
Duration of sedation | During ICU stay. Expected average 21 days
  Duration of sedation during ICU stay in days
ICU LOS | During ICU stay. Up to 30 days
  Length of ICU stay in days
Hospital Mortality | 90 days
  Hospital LOS in days
Physical function | ICU discharge (baseline) and change from baseline at 3 months
  Measure of handgrip strength though a high precision dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, MA, PhD, Study Chair — DIRECTOR ICU
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wunsch H, Angus DC, Harrison DA, Collange O, Fowler R, Hoste EA, de Keizer NF, Kersten A, Linde-Zwirble WT, Sandiumenge A, Rowan KM. Variation in critical care services across North America and Western Europe. Crit Care Med. 2008 Oct;36(10):2787-93, e1-9. doi: 10.1097/CCM.0b013e318186aec8. PMID 18766102
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] 4. Torres J, Veiga C, Pinto F, et al. Post intensive care syndrome- from risk at ICU admission to 3 months follow-up clinic. Intensive Care Med Experimental 2015, 3 (Suppl 1): A448.
- [Background] 5. Ramnarain D, Rutten A, Van der Nat G, et al. The impact of post intensive care syndrome in patients surviving the ICU: the downside of ICU treatment. Intensive Care Med Experimental 2015, 3 (Suppl 1): A530.
- [Background] de Azevedo JR, Montenegro WS, Rodrigues DP, de C Souza SC, Araujo VF, de Paula MP, Prazeres PH, da Luz Leitao A, Mendonca AV. Long-term cognitive outcomes among unselected ventilated and non-ventilated ICU patients. J Intensive Care. 2017 Feb 17;5:18. doi: 10.1186/s40560-017-0213-4. eCollection 2017. PMID 28239475
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258